CLINICAL TRIAL: NCT04342455
Title: Evaluation the Diagnostic Efficacy of a Low-dose Radiation and Contrast Agent Exposure Protocol for Coronary Computed Tomography Angiography(CTA)on Coronary Artery Disease in Diabetic Patients
Brief Title: A Low-dose Radiation and Contrast Agent Exposure Protocol for Coronary CTA in Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Yangtze River Pharmaceutical Group Co., Ltd. (Industry); Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: XJTU1AF2018LSY-23
Record Dates: First submitted 2018-09-05; First posted 2020-04-13 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-03

CONDITIONS: Coronary Artery Disease
Keywords: Coronary CT angiography; Iodixanol; Diabetes; Diagnosis
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus; Disease

STUDY DESIGN:
Intervention Model Description: All subjects undergo coronary CTA and invasive coronary angiography (ICA), but coronary CTA examinees are divided into two groups performing different scanning and contrast protocols.
Who Masked: Participant, Outcomes Assessor
Masking Description: This study belongs to a diagnostic test of CT angiography . All participants use the same contrast agent. The interventions on the two groups are different in scanning protocol of CTA. The examinees and image readers are blind, and the scanning technician is unblinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional scanning protocol group (No Intervention): In coronary CTA examination,each subject will be injected 50 ml contrast agent (Iodixanol 320) with the flow rate of 5 ml/s in tube voltage of 120 kVp.
- double-low scanning protocol group (Experimental): In coronary CTA examination,the tube voltage(70，80,100kVp),contrast agent(Iodixanol 320) volume and flow rate of each subject are adapted to his or her cardiac ejection fraction(EF) and body mass index(BMI).
  Interventions: Other: double-low scanning

INTERVENTIONS:
Other: double-low scanning — a CT angiography protocol with low radiation and contrast agent exposure
  Arms: double-low scanning protocol group

SUMMARY:
To assess diagnostic accuracy,image quality and renal safety of a double low-dose coronary CTA protocol at coronary artery evaluation in patients with diabetes by using invasive coronary angiography(ICA) as the reference method and to compare the results with those obtained traditional dose protocol. The study will randomly include about 400 consecutive participants aged 18 to 80 years old who had been diagnosed with diabetes and suspected coronary artery disease.All participants undergo ICA and coronary CT angiography performed with a whole-heart CT scan.Coronary segment interpretability,image quality based on a four-point Likert scale,blood indicators of renal function will be accessed between double low-dose CTA protocol and traditional CTA protocol. Investigators hypothesize that an individualized coronary CTA protocol that appropriately reduces radiation dose and contrast dose does not affect image quality and diagnostic accuracy, and can reduce the risk of kidney damage in high-risk patients.

DETAILED DESCRIPTION:
The study has been approved by the local ethics committee and allparticipants will be provided written informed consent. Iodixanol 320 mg/ml is injected followed by 30 ml of saline solution.In the test group,the tube voltage,contrast agent volume and flow rate are adapted to cardiac ejection fraction(EF) and body mass index(BMI)according to the pretest. participants in the contract group are injected 50 ml contrast agent with the flow rate of 5 ml/s in tube voltage of 120 kVp. All participants are scanned in automatic tube current.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years old and ≤ 80 years old;
* patients who have previously diagnosed diabetes;
* patients with suspected coronary artery disease and undergoing coronary CT angiography (CTA);
* Subjects are fully informed and provided written informed consent.

Exclusion Criteria:

* The exclusion criteria are pregnancy and lactation women or recent birth planners
* patients with Iodine contrast agent contraindications (such as a history of severe allergy history with iodine contrast agents, hyperthyroidism, etc.)
* patients with chronic kidney disease (Phase 4-5, eGFR <30 ml/min/1.73 m2)
* patients who have undergone coronary stent implantation or coronary artery bypass surgery
* patients who have received iodine contrast-related tests within 24 hours
* participated in other clinical trials within 3 months
* other circumstances that the investigator believes are not suitable for participation in the trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-10-07 (Actual); Primary Completion 2020-09-15 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
diagnosis accuracy (including sensitivity,specificity of the low-dose radiation and contrast agent exposure protocol for coronary CTA) | three years
  Comparing with invasive coronary angiography,if the low-dose radiation and contrast agent exposure protocol for coronary CTA can detect significant（>50%）stenosis.

SECONDARY OUTCOMES:
image quality | three years
  two independent blinded readers semi-quantitatively the image quality.Compare the difference in image quality score between the the low-dose radiation and contrast agent exposure protocol and the traditional protocol.
image quality | three years
  Compare the difference in signal-to-noise ratio (SNR),contrast-to-noise ratio (CNR) and Contrast density between the two groups.
kidney function | three years
  Compare the difference in the level of creatinine(Cr) and cystatin C in serum between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Jian, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China